CLINICAL TRIAL: NCT00602472
Title: A Randomised, Double-blind, Placebo-controlled Parallel Group Efficacy and Safety Study of BI 1356 (5 mg) Administered Orally Once Daily Over 24 Weeks, With an Open-label Extension to One Year (Placebo Patients Switched to BI 1356), in Type 2 Diabetic Patients With Insufficient Glycaemic Control Despite a Therapy of Metformin in Combination With a Sulphonylurea
Brief Title: BI 1356 (Linagliptin) in Combination With Metformin and a Sulphonylurea in Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1218.18; 2007-002450-28 (EudraCT Number: EudraCT)
Record Dates: First submitted 2008-01-15; First posted 2008-01-28 (Estimated); Results first posted 2011-06-15 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Linagliptin

ARMS (2):
- linagliptin 5 mg (Experimental): linagliptin 5 mg once daily
  Interventions: Drug: linagliptin
- placebo (Placebo Comparator): placebo matching linagliptin 5 mg tablets
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: linagliptin — active
  Arms: linagliptin 5 mg
Drug: placebo — placebo to linagliptin 5 mg
  Arms: placebo

SUMMARY:
The objective of the current study is to investigate the efficacy, safety and tolerability of BI 1356 (5 mg once daily) compared to placebo given for 24 weeks as add-on therapy to metformin in combination with a sulphonylurea in patients with type 2 diabetes mellitus with insufficient glycaemic control.

ELIGIBILITY:
Inclusion criteria:

1. Male and female patients with a diagnosis of type 2 diabetes mellitus, currently treated only with a stable total daily dose of preferably* >/= 1500 mg metformin and a dose of a sulphonylurea drug that has been documented, by the Investigator, to be the individual maximum tolerated dose of that sulphonylurea drug. Both the dose and dosing regimen of metformin and the sulphonylurea must be stable (i.e. unchanged) for 10 weeks prior to informed consent, and must not be changed for the duration of the trial
2. Glycosylated haemoglobin A1 (HbA1c) >/= 7.0 and </= 10.0% at the screening Visit 1a and at Visit 2 (start of placebo run-in phase)
3. Age >/= 18 and </= 80 years at Visit 1a (screening)
4. BMI (Body Mass Index) </= 40 kg/m2 at Visit 1a (screening)
5. Signed and dated written informed consent, at the latest by the date of Visit 1a, in accordance with GCP and local legislation *Patients currently treated with a total daily dose of less than 1500 mg metformin can be included in the trial if the Investigator has documented that the dose is the maximum tolerated dose of metformin for that patient.

Exclusion criteria:

1. Myocardial infarction, stroke or TIA (transient ischaemic attack) within 6 months prior to the date of informed consent
2. Impaired hepatic function, defined by serum levels of either alanine transaminase (ALT/SGPT), aspartase transaminase (AST/SGOT), or alkaline phosphatase (ALP) above 3 times the upper limit of normal (ULN), as determined at Visit 1a
3. Renal failure or renal impairment (serum creatinine >/= 1.5 mg/dl) as determined at Visit 1a
4. Treatment with rosiglitazone or pioglitazone within 3 months prior to the date of informed consent
5. Treatment with GLP-1 analogues (e.g. exenatide) within 3 months prior to the date of informed consent
6. Treatment with insulin within 3 months prior to the date of informed consent
7. Treatment with anti-obesity drugs (e.g. sibutramine, rimonabant, orlistat) within 3 months prior to the date of informed consent
8. Current treatment with systemic steroids (i.e. at the time of informed consent) or a change in the dosage of thyroid hormones within 6 weeks prior to the date of informed consent
9. Pre-menopausal women (last menstruation </= 1 year prior to the date of informed consent) who:

   * are nursing or pregnant
   * or are of child-bearing potential and are not practicing an acceptable method of birth control, or do not plan to continue using this method throughout the study and do not agree to periodic pregnancy testing during their participation in the trial. Acceptable methods of birth control include transdermal patch, intra uterine devices/systems (IUDs/IUSs), oral, implantable or injectable contraceptives, sexual abstinence and vasectomised partner. No exception will be made.
10. Known hypersensitivity or allergy to the investigational product or its excipients or to the trial background therapy (i.e. metformin in combination with a sulphonylurea) or sulphonamides
11. Dehydration (as confirmed by the Investigators clinical opinion)
12. Current acute or chronic metabolic acidosis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1058 (Actual)
Dates: Start 2008-02; Primary Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (100):
- Argentina (14):
  - 1218.18.54001 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1218.18.54002 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1218.18.54004 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1218.18.54005 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1218.18.54010 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1218.18.54014 Boehringer Ingelheim Investigational Site, Corrientes
  - 1218.18.54009 Boehringer Ingelheim Investigational Site, Córdoba
  - 1218.18.54013 Boehringer Ingelheim Investigational Site, Córdoba
  - 1218.18.54003 Boehringer Ingelheim Investigational Site, Mar del Plata
  - 1218.18.54012 Boehringer Ingelheim Investigational Site, Mar del Plata
  - 1218.18.54011 Boehringer Ingelheim Investigational Site, Mendoza
  - 1218.18.54015 Boehringer Ingelheim Investigational Site, Parque Velez Sarfield
  - 1218.18.54006 Boehringer Ingelheim Investigational Site, Rosario
  - 1218.18.54007 Boehringer Ingelheim Investigational Site, Salta
- Belgium (7):
  - 1218.18.32005 Boehringer Ingelheim Investigational Site, Bruges
  - 1218.18.32007 Boehringer Ingelheim Investigational Site, Brussels
  - 1218.18.32006 Boehringer Ingelheim Investigational Site, Edegem
  - 1218.18.32004 Boehringer Ingelheim Investigational Site, Genk
  - 1218.18.32003 Boehringer Ingelheim Investigational Site, Ghent
  - 1218.18.32002 Boehringer Ingelheim Investigational Site, Huy
  - 1218.18.32001 Boehringer Ingelheim Investigational Site, Liège
- Canada (12):
  - 1218.18.01005 Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - 1218.18.01010 Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - 1218.18.01003 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1218.18.01011 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1218.18.01006 Boehringer Ingelheim Investigational Site, Etobicoke, Ontario
  - 1218.18.01009 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1218.18.01002 Boehringer Ingelheim Investigational Site, London, Ontario
  - 1218.18.01012 Boehringer Ingelheim Investigational Site, Oakville, Ontario
  - 1218.18.01008 Boehringer Ingelheim Investigational Site, Sarnia, Ontario
  - 1218.18.01001 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1218.18.01004 Boehringer Ingelheim Investigational Site, Montague, Prince Edward Island
  - 1218.18.01007 Boehringer Ingelheim Investigational Site, Saskatoon, Saskatchewan
- China (15):
  - 1218.18.86001 Boehringer Ingelheim Investigational Site, Beijing
  - 1218.18.86002 Boehringer Ingelheim Investigational Site, Beijing
  - 1218.18.86004 Boehringer Ingelheim Investigational Site, Beijing
  - 1218.18.86013 Boehringer Ingelheim Investigational Site, Chengdu, Sichuan Province
  - 1218.18.86009 Boehringer Ingelheim Investigational Site, Dalian
  - 1218.18.86011 Boehringer Ingelheim Investigational Site, Guangzhou
  - 1218.18.86014 Boehringer Ingelheim Investigational Site, Haerbin
  - 1218.18.86005 Boehringer Ingelheim Investigational Site, Nanjing, Jiangsu Province
  - 1218.18.86008 Boehringer Ingelheim Investigational Site, Qingdao
  - 1218.18.86015 Boehringer Ingelheim Investigational Site, Shanghai
  - 1218.18.86010 Boehringer Ingelheim Investigational Site, Shenyang
  - 1218.18.86003 Boehringer Ingelheim Investigational Site, Weizikeng
  - 1218.18.86007 Boehringer Ingelheim Investigational Site, Wuhan
  - 1218.18.86012 Boehringer Ingelheim Investigational Site, Wuhan, Hubei Province
  - 1218.18.86006 Boehringer Ingelheim Investigational Site, Xian, Shanxi Province
- Germany (9):
  - 1218.18.49004 Boehringer Ingelheim Investigational Site, Aschaffenburg
  - 1218.18.49028 Boehringer Ingelheim Investigational Site, Bad Mergentheim
  - 1218.18.49022 Boehringer Ingelheim Investigational Site, Berlin
  - 1218.18.49024 Boehringer Ingelheim Investigational Site, Bosenheim
  - 1218.18.49020 Boehringer Ingelheim Investigational Site, Dresden
  - 1218.18.49101 Boehringer Ingelheim Investigational Site, Mainz
  - 1218.18.49003 Boehringer Ingelheim Investigational Site, Neuwied
  - 1218.18.49007 Boehringer Ingelheim Investigational Site, Nuremberg
  - 1218.18.49014 Boehringer Ingelheim Investigational Site, Saarbrücken
- Philippines (5):
  - 1218.18.63005 Boehringer Ingelheim Investigational Site, Manila
  - 1218.18.63002 Boehringer Ingelheim Investigational Site, Marikina City
  - 1218.18.63001 Boehringer Ingelheim Investigational Site, Pasig
  - 1218.18.63004 Boehringer Ingelheim Investigational Site, Quezon City
  - 1218.18.63003 Boehringer Ingelheim Investigational Site, San Juan City
- Russia (5):
  - 1218.18.70014 Boehringer Ingelheim Investigational Site, Arkhangelsk
  - 1218.18.70012 Boehringer Ingelheim Investigational Site, Moscow
  - 1218.18.70013 Boehringer Ingelheim Investigational Site, Rostov-on-Don
  - 1218.18.70015 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1218.18.70016 Boehringer Ingelheim Investigational Site, Samara
- South Korea (11):
  - 1218.18.82004 Boehringer Ingelheim Investigational Site, Busan
  - 1218.18.82011 Boehringer Ingelheim Investigational Site, Daegu
  - 1218.18.82008 Boehringer Ingelheim Investigational Site, Incheon
  - 1218.18.82010 Boehringer Ingelheim Investigational Site, Jeonju
  - 1218.18.82002 Boehringer Ingelheim Investigational Site, Pusan
  - 1218.18.82001 Boehringer Ingelheim Investigational Site, Seoul
  - 1218.18.82005 Boehringer Ingelheim Investigational Site, Seoul
  - 1218.18.82006 Boehringer Ingelheim Investigational Site, Seoul
  - 1218.18.82007 Boehringer Ingelheim Investigational Site, Seoul
  - 1218.18.82009 Boehringer Ingelheim Investigational Site, Seoul
  - 1218.18.82003 Boehringer Ingelheim Investigational Site, Suwon
- Taiwan (8):
  - 1218.18.88605 Boehringer Ingelheim Investigational Site, Changhua
  - 1218.18.88604 Boehringer Ingelheim Investigational Site, Taichung
  - 1218.18.88606 Boehringer Ingelheim Investigational Site, Tainan
  - 1218.18.88601 Boehringer Ingelheim Investigational Site, Taipei
  - 1218.18.88602 Boehringer Ingelheim Investigational Site, Taipei
  - 1218.18.88603 Boehringer Ingelheim Investigational Site, Taipei
  - 1218.18.88607 Boehringer Ingelheim Investigational Site, Taipei
  - 1218.18.88608 Boehringer Ingelheim Investigational Site, Taoyuan District
- Turkey (Türkiye) (4):
  - 1218.18.90003 Boehringer Ingelheim Investigational Site, Erzurum
  - 1218.18.90005 Boehringer Ingelheim Investigational Site, Istanbul
  - 1218.18.90001 Boehringer Ingelheim Investigational Site, Izmir
  - 1218.18.90004 Boehringer Ingelheim Investigational Site, Konya
- United Kingdom (10):
  - 1218.18.44005 Boehringer Ingelheim Investigational Site, Ashford
  - 1218.18.44004 Boehringer Ingelheim Investigational Site, Baillieston, Glasgow
  - 1218.18.44001 Boehringer Ingelheim Investigational Site, Bath
  - 1218.18.44003 Boehringer Ingelheim Investigational Site, Burbage
  - 1218.18.44010 Boehringer Ingelheim Investigational Site, Bury Saint Edmonds
  - 1218.18.44009 Boehringer Ingelheim Investigational Site, Cardiff
  - 1218.18.44008 Boehringer Ingelheim Investigational Site, Glasgow
  - 1218.18.44002 Boehringer Ingelheim Investigational Site, Penarth
  - 1218.18.44006 Boehringer Ingelheim Investigational Site, Reading
  - 1218.18.44007 Boehringer Ingelheim Investigational Site, Waterloo, Liverpool

REFERENCES:
- [Derived] Del Prato S, Patel S, Crowe S, von Eynatten M. Efficacy and safety of linagliptin according to patient baseline characteristics: A pooled analysis of three phase 3 trials. Nutr Metab Cardiovasc Dis. 2016 Oct;26(10):886-92. doi: 10.1016/j.numecd.2016.06.015. Epub 2016 Jul 1. PMID 27484756
- [Derived] Zeng Z, Yang JK, Tong N, Yan S, Zhang X, Gong Y, Woerle HJ. Efficacy and safety of linagliptin added to metformin and sulphonylurea in Chinese patients with type 2 diabetes: a sub-analysis of data from a randomised clinical trial. Curr Med Res Opin. 2013 Aug;29(8):921-9. doi: 10.1185/03007995.2013.805123. Epub 2013 Jun 4. PMID 23672632
- [Derived] Johansen OE, Neubacher D, von Eynatten M, Patel S, Woerle HJ. Cardiovascular safety with linagliptin in patients with type 2 diabetes mellitus: a pre-specified, prospective, and adjudicated meta-analysis of a phase 3 programme. Cardiovasc Diabetol. 2012 Jan 10;11:3. doi: 10.1186/1475-2840-11-3. PMID 22234149
- [Derived] Owens DR, Swallow R, Dugi KA, Woerle HJ. Efficacy and safety of linagliptin in persons with type 2 diabetes inadequately controlled by a combination of metformin and sulphonylurea: a 24-week randomized study. Diabet Med. 2011 Nov;28(11):1352-61. doi: 10.1111/j.1464-5491.2011.03387.x. PMID 21781152

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Patients randomized to receive treatment with matching placebo
- Linagliptin: Patients randomized to receive treatment with Linagliptin 5mg
Period: Overall Study
Arm/Group | Placebo | Linagliptin
Started | 263 (3 randomised patients never took medication.) | 792 (3 randomised patients never took medication.)
Completed | 242 (number who completed treatment) | 734 (number who completed treatment)
Not Completed | 21 | 58
Not completed — Adverse Event | 5 | 23
Not completed — Protocol Violation | 4 | 19
Not completed — Withdrawal by Subject | 8 | 14
Not completed — Other incl. lack of efficacy | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Linagliptin | Total
Number analyzed (Participants) | 263 | 792 | 1055
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.6 (9.7) | 58.3 (9.9) | 58.1 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136 | 421 | 557
  Male | 127 | 371 | 498
Body mass index (BMI) continuous [Mean (Standard Deviation); unit: kg/m^2] | 28.16 (4.52) | 28.38 (4.79) | 28.33 (4.72)
Glycosylated Hemoglobin A1 (HbA1c) [Mean (Standard Deviation); unit: Percent] | 8.14 (0.84) | 8.15 (0.80) | 8.14 (0.81)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] | 162.6 (37.1) | 159.3 (36.5) | 160.1 (36.6)

OUTCOME MEASURES:

1. Primary Outcome: HbA1c Change From Baseline to Week 24
Description: HbA1c is measured as a percentage. Thus, this change from baseline reflects the Week 24 HbA1c percent minus the baseline HbA1c percent. Means are treatment adjusted for baseline HbA1c and previous anti-diabetic medication.
Time Frame: Baseline and week 24
Population: The Full Analysis Set (FAS) included all treated and randomised patients with a baseline and at least one on treatment HbA1c measurement available. Last observation carried forward (LOCF) was used as the imputation rule.
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 262 | 778
Percent | -0.10 (0.05) | -0.72 (0.03)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin; Linagliptin vs. Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.62, 95% CI [-0.73 to -0.50], Standard Error of Mean 0.06

2. Secondary Outcome: HbA1c Change From Baseline to Week 6
Description: HbA1c is measured as a percentage. Thus, this change from baseline reflects the Week 6 HbA1c percent minus the baseline HbA1c percent. Means are treatment adjusted for baseline HbA1c and previous anti-diabetic medication.
Time Frame: Baseline and week 6
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 262 | 778
Percent | -0.18 (0.03) | -0.67 (0.02)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin; Linagliptin vs. Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.49, 95% CI [-0.56 to -0.41], Standard Error of Mean 0.04

3. Secondary Outcome: HbA1c Change From Baseline to Week 12
Description: HbA1c is measured as a percentage. Thus, this change from baseline reflects the Week 12 HbA1c percent minus the baseline HbA1c percent. Means are treatment adjusted for baseline HbA1c and previous anti-diabetic medication.
Time Frame: Baseline and week 12
Population: The Full Analysis Set (FAS) included all treated and randomised patients with a baseline and at least one on-treatment.
  HbA1c measurement available. Last observation carried forward (LOCF) was used as the imputation rule.
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 262 | 778
Percent | -0.15 (0.04) | -0.84 (0.03)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin; Linagliptin vs. Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.68, 95% CI [-0.78 to -0.58], Standard Error of Mean 0.05

4. Secondary Outcome: HbA1c Change From Baseline to Week 18
Description: HbA1c is measured as a percentage. Thus, this change from baseline reflects the Week 18 HbA1c percent minus the baseline HbA1c percent. Means are treatment adjusted for baseline HbA1c and previous anti-diabetic medication.
Time Frame: Baseline and week 18
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 262 | 778
Percent | -0.11 (0.05) | -0.81 (0.03)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin; Linagliptin vs. Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.69, 95% CI [-0.80 to -0.59], Standard Error of Mean 0.05

5. Secondary Outcome: FPG Change From Baseline to Week 24
Description: This change from baseline reflects the Week 24 FPG minus the baseline FPG. Means are treatment-adjusted for baseline HbA1c, baseline FPG and previous anti-diabetic medication.
Time Frame: Baseline and week 24
Population: This population includes the FAS using the LOCF imputation, with the further restriction of patients with a baseline and post-baseline FPG value.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 248 | 739
mg/dL | 8.1 (2.4) | -4.6 (1.4)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin; Linagliptin vs. Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -12.7, 95% CI [-18.1 to -7.3], Standard Error of Mean 2.8

6. Secondary Outcome: FPG Change From Baseline to Week 6
Description: This change from baseline reflects the Week 6 FPG minus the baseline FPG. Means are treatment-adjusted for baseline HbA1c, baseline FPG and previous anti-diabetic medication.
Time Frame: Baseline and week 6
Population: as for outcome 5
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 248 | 739
mg/dL | 6.3 (2.0) | -11.5 (1.2)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin; Linagliptin vs. Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -17.8, 95% CI [-22.4 to -13.2], Standard Error of Mean 2.3

7. Secondary Outcome: FPG Change From Baseline to Week 12
Description: This change from baseline reflects the Week 12 FPG minus the baseline FPG. Means are treatment adjusted for baseline HbA1c, baseline FPG and previous anti-diabetic medication.
Time Frame: Baseline and week 12
Population: as for outcome 5
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 248 | 739
mg/dL | 6.2 (2.0) | -9.5 (1.2)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin; Linagliptin vs. Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -15.7, 95% CI [-20.3 to -11.1], Standard Error of Mean 2.4

8. Secondary Outcome: FPG Change From Baseline to Week 18
Description: This change from baseline reflects the Week 18 FPG minus the Week 0 FPG. Means are treatment-adjusted for baseline HbA1c, baseline FPG and previous anti-diabetic medication
Time Frame: Baseline and week 18
Population: as for outcome 5
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 248 | 739
mg/dL | 7.4 (2.2) | -4.7 (1.3)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin; Linagliptin vs. Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -12.1, 95% CI [-17.2 to -7.1], Standard Error of Mean 2.6

9. Secondary Outcome: Percentage of Patients With HbA1c <7.0% at Week 24
Description: The percentage of patients with an HbA1c value below 7% at week 24 was calculated for each treatment arm. If a patient did not have an HbA1c value at week 24 they were considered a failure, so HbA1c above 7%. Only patients with baseline HbA1c >= 7%
Time Frame: Baseline and week 24
Population: This population includes the FAS with baseline HbA1c >= 7.0%. Non-completers were considered as failure imputation (NCF).
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 247 | 742
percentage of patients | 8.1 (0) | 29.2 (0)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin; Linagliptin vs. Placebo The odds-ratio is based on a logistic regression model including baseline HbA1c and previous antidiabetes medication; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 5.510, 95% CI [3.332 to 9.111]

10. Secondary Outcome: Percentage of Patients With HbA1c < 7.0% at Week 24
Description: The percentage of patients with an HbA1c value below 7% at week 24 was calculated for each treatment arm. If a patient did not have an HbA1c value at week 24 they were considered a failure, so HbA1c above 7%.
Time Frame: Baseline and week 24
Population: This population includes the Full Analysis Set (FAS). Non-completers were considered as failure imputation (NCF).
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 262 | 778
percentage of patients | 9.2 | 31.2

11. Secondary Outcome: Percentage of Patients With HbA1c <6.5% at Week 24
Description: The percentage of patients with an HbA1c value below 6.5% at week 24 was calculated for each treatment arm. If a patient did not have an HbA1c value at week 24 they were considered a failure, so HbA1c above 6.5%. Only patients with baseline HbA1c >= 6.5%
Time Frame: Baseline and week 24
Population: This population includes the FAS with baseline HbA1c >= 6.5%. Non-completers were considered as failure imputation (NCF).
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 262 | 777
percentage of patients | 4.2 (0) | 13.1 (0)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 3.818, 95% CI [1.989 to 7.327]

12. Secondary Outcome: Percentage of Patients With HbA1c<6.5% at Week 24
Description: The percentage of patients with an HbA1c value below 6.5% at week 24 was calculated for each treatment arm. If a patient did not have an HbA1c value at week 24 they were considered a failure, so HbA1c above 6.5%
Time Frame: Baseline and week 24
Population: This population includes the Full Analysis Set (FAS). Non-completers were considered as failure imputation (NCF).
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 262 | 778
percentage of patients | 4.2 | 13.1

13. Secondary Outcome: Percentage of Patients Who Have a HbA1c Lowering by 0.5% at Week 24
Description: The percentage of patients with an HbA1c reduction greater than 0.5% at week 24 from baseline was calculated for each treatment arm. If a patient did not have an HbA1c value at week 24 they were considered a failure, so HbA1c reduction less than 0.5%
Time Frame: Baseline and week 24
Population: The Full Analysis Set (FAS) included all patients with a baseline and at least one on treatment HbA1c measurement available. Non-completers were considered as failure imputation (NCF).
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 262 | 778
percentage of patients | 30.2 (0) | 58.2 (0)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 3.360, 95% CI [2.474 to 4.562]

ADVERSE EVENTS:
Time Frame: From day of first drug dose until 7 days after last dose, with an average of 166 days
Arm/Group | Placebo | Linagliptin
Serious Adverse Events (participants affected / at risk) | 10/263 | 25/792
Other Adverse Events (participants affected / at risk) | 94/263 | 273/792
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=263) | Linagliptin (N=792)
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 1
Angina unstable (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Myocarditis (Cardiac disorders) | 0 | 1
Eye swelling (Eye disorders) | 0 | 1
Glaucoma (Eye disorders) | 1 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1
Vitreous haemorrhage (Eye disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Gingival swelling (Gastrointestinal disorders) | 0 | 1
Lip swelling (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Chest discomfort (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Otitis media chronic (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 1 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1
Tension headache (Nervous system disorders) | 0 | 1
Ketonuria (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1
Urinary bladder polyp (Renal and urinary disorders) | 1 | 0
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 1
Hypertensive crisis (Vascular disorders) | 0 | 2
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=263) | Linagliptin (N=792)
Nasopharyngitis (Infections and infestations) | 12 | 41
Upper respiratory tract infection (Infections and infestations) | 24 | 46
Urinary tract infection (Infections and infestations) | 14 | 25
Hyperglycaemia (Metabolism and nutrition disorders) | 23 | 44
Hypoglycaemia (Metabolism and nutrition disorders) | 39 | 180

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.